CLINICAL TRIAL: NCT01231919
Title: A Phase I Study of MK-2206, an AKT Inhibitor, in Pediatric Patients With Recurrent or Refractory Solid Tumors or Leukemia
Brief Title: MK2206 in Treating Younger Patients With Recurrent or Refractory Solid Tumors or Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02612; NCI-2011-02612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687929; COG-ADVL1013; ADVL1013 (Other: COG Phase I Consortium); ADVL1013 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Leukemias of Ambiguous Lineage; Acute Myeloid Leukemia/Transient Myeloproliferative Disorder; Acute Undifferentiated Leukemia; Aggressive NK-cell Leukemia; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Blastic Plasmacytoid Dendritic Cell Neoplasm; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Intraocular Lymphoma; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Myeloid/NK-cell Acute Leukemia; Noncutaneous Extranodal Lymphoma; Post-transplant Lymphoproliferative Disorder; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Myeloproliferative Syndrome, Transient; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Blastic Plasmacytoid Dendritic Cell Neoplasm; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor) (Experimental): Patients receive oral Akt inhibitor MK2206 every other day (schedule 1) OR once weekly (schedule 2) on days 1-28. Treatment repeats every 28 days for up 12 courses (1 year) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt inhibitor MK2206; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: diagnostic laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects, best way to give, and best dose of Akt inhibitor MK2206 (MK2206) in treating patients with recurrent or refractory solid tumors or leukemia. MK2206 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To estimate the maximum-tolerated dose (MTD) and/or recommended phase 2 dose of MK-2206 (Akt inhibitor MK2206) administered orally every other day (schedule 1) or once weekly (schedule 2) to children with refractory or recurrent solid malignancies, including central nervous system (CNS) tumors or lymphomas.

II. To define and describe the toxicities of MK-2206 in children with refractory solid malignancies administered on this schedule.

III. To assess the tolerability of MK-2206 at the solid tumor MTD in patients with recurrent or refractory leukemia.

IV. To characterize the pharmacokinetics of MK-2206 in children with recurrent or refractory cancer. (exploratory)

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of MK-2206 within the confines of a phase 1 study.(exploratory) II. To evaluate biological activity of MK-2206 by measuring phosphatidylinositol 3 kinase (PI3K)/protein kinase B (AKT)/mammalian target of rapamycin (mTOR) signaling in tumor and peripheral blood mononuclear cells and measure the expression of biomarkers related to AKT activation phenotypes. (exploratory)

OUTLINE: This is a dose-escalation study (part A) followed by treatment at the maximum-tolerated dose (part B).

Patients receive Akt inhibitor MK2206 orally (PO) every other day (schedule 1) OR once weekly (schedule 2) on days 1-28. Treatment repeats every 28 days for up 12 courses (1 year) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area > 0.5 m^2 when enrolling on dose levels 0 or 1 of the every other day schedule; no body surface area (BSA) restrictions apply to patients enrolling on higher dose levels; no BSA restrictions apply to patients enrolling on any dose level of the weekly schedule.
* Diagnosis:

  * Part A (both schedules): Patients must have a diagnosis of recurrent or refractory solid tumors, including central nervous system (CNS) tumors or lymphoma; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
  * Part B (both schedules): Patients must have a diagnosis of recurrent or refractory leukemia
* Disease status:

  * Solid tumors: Patients must have either measurable or evaluable disease
  * Leukemia: Patients must have >= 5% blasts in the bone marrow; active extramedullary disease (except for leptomeningeal disease) may also be present
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; note: neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 1 week prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy
* Myelosuppressive chemotherapy:

  * Solid tumors: Patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
  * Leukemia:

    * Patients with leukemia who relapse while receiving standard maintenance chemotherapy will not be required to have a waiting period before enrollment onto this study
    * Patients who relapse while they are not receiving standard maintenance therapy, must have fully recovered from all acute toxic effects of prior therapy. At least 14 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea
    * Note: Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of MK-2206
* At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines
* At least 3 half-lives of the antibody after the last dose of a monoclonal antibody
* >= 2 weeks for local palliative radiation therapy (XRT) (small port); >= 24 weeks must have elapsed if prior total body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* Stem cell infusion without TBI: No evidence of active graft vs. host disease and >= 8 weeks must have elapsed since transplant or stem cell infusion
* Bone marrow transplantation: >= 3 months prior to study enrollment
* For patients with solid tumors without known bone marrow involvement including patients who are status post stem cell transplantation:
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* For patients with solid tumors with known bone marrow metastatic disease:
* These patients are eligible for study provided they meet the blood count criteria and are not known to be refractory to red cell or platelet transfusions; note: these patients are not evaluable for hematologic toxicity
* For patients with leukemia (Part B):
* Blood counts are not required to be normal prior to enrollment on this trial; however, platelet count has to be >= 20,000/mm^3 (may receive platelet transfusions)
* Creatinine clearance or radioisotope GFR >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Patients with solid tumors:

  * Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
  * Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
  * Serum albumin >= 2 g/dL
* Patients with leukemias:

  * Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) =< 225 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
  * Serum albumin >= 2 g/dL
* Corrected QT interval (QTc) =< 450 msec
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] v4) resulting from prior therapy must be =< grade 2
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Slides or tissue blocks from either initial diagnosis or relapse must be available for central review; tissue blocks or slides must be sent; if tissue blocks or slides are unavailable, the study chair must be notified prior to study enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anticancer agents are not eligible [except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy]; patients with leukemia may receive intrathecal therapy
* Patients must not be receiving enzyme-inducing anticonvulsants
* Patients receiving insulin or growth hormone therapy are not eligible
* Patients on medications that may cause corrected QT (QTc) interval prolongation are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post transplant are not eligible for this trial
* Patients must be able to swallow whole tablets; nasogastric or G tube administration is not allowed
* Patients who have an uncontrolled infection are not eligible
* Patients with known type I or type II diabetes mellitus are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
MTD and/or recommended phase 2 dose of Akt inhibitor MK2206 determined according to incidence of dose-limiting toxicities (DLTs) graded using CTCAE v4.0 (Part A) | 28 days
  The MTD will be the maximum dose at which fewer than one-third of patients experience DLT during course 1 of therapy.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of Akt inhibitor MK-2206 | Baseline, 0.5, 1.5, 3, 6-8, 24, 48 hours day 1 course 1; pre-dose and 6-8 hours post-dose (optional) day 15 (Schedule 1); baseline, 0.5, 1.5, 3, 6-8, 24, 48 hours day 1 course 1; pre-dose days 8 and 15; 6-8 hours post-dose day 15 (optional) (Schedule 2)
  Summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Antitumor activity assessed by Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 | Up to 30 days
Levels of activation of downstream signaling molecules | Up to day 15 of course 1
  Summarized using descriptive statistics at each timepoint. The Wilcoxon signed-rank test or Friedman's test may be used as a preliminary test of change in activity over two or more timepoints.
Mutations or amplification of upstream signaling molecules | Baseline
  Summarized using descriptive statistics at each timepoint. The Wilcoxon signed-rank test or Friedman's test may be used as a preliminary test of change in activity over two or more timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — COG Phase I Consortium
Locations (25):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mark O Hatfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec